CLINICAL TRIAL: NCT00266370
Title: A Pathology Reference Laboratory for the Study of Infectious Diseases and Malignant Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Other Study IDs: CL-094-CP-01
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2005-12-19 (Estimated); Status verified 2005-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
1. To establish a pathology reference laboratory for the consultation on the diagnosis of infectious diseases and lymphoma.
2. To study the specific pathogens on 100 cases of unexplained death due to infectious diseases in the files of Taiwan CDC and the Forensic Institutes of Department of Law and Justice.
3. To study the distribution of children lymphoid lesions in Vietnam and Taiwan and their virus association.
4. To establish a tissue bank for infectious diseases and lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of infectious diseases and lymphoma.

Exclusion Criteria:

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2009-12

CONTACTS AND LOCATIONS:
Overall Officials: Ih-Jen Su, M.D., Ph.D., Principal Investigator — Division of Clinical Research, National Health Research Institutes
Locations (1):
- National Health Research Institutes, Zhunan Town, Miaoli County, Taiwan